CLINICAL TRIAL: NCT06181968
Title: Echocardiography and Lung Ultrasound Combined Into a Rapid Cardiothoracic Ultrasound Protocol (CaTUS) for Guiding Decongestive Treartment on a Day-to-day Basis in Patients Hospitalized for Acute Heart Failure With Pulmonary Congestion
Brief Title: Ultrasound-guided Treatment in Acute Heart Failure
Acronym: ECHO-AHF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI not workining at KUH anymore.
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Juha Hartikainen, Clinical Professor, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KUH5101120
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Acute Heart Failure; Congestion
Keywords: Acute Heart Failure; Echocardiography; Lung Ultrasound

STUDY DESIGN:
Intervention Model Description: Randomized controlled, blinded
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the treating physician on the ward will know which arm the patient belongs to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Active Comparator): Congestive therapy will be guided by findings on daily cardiac- and lung ultrasound
  Interventions: Diagnostic Test: Cardiothoracic ultrasound protocol
- Control Arm (Sham Comparator): This arm will have the same ultrasound exams done daily as the treatment arm, but information will not be available for the treating physician for guiding therapy
  Interventions: Diagnostic Test: Cardiothoracic ultrasound protocol

INTERVENTIONS:
Diagnostic Test: Cardiothoracic ultrasound protocol — Combined echocardiography and lung ultrasound for guiding therapy

SUMMARY:
A randomized non-blinded study comparing ultrasound-guided therapy with conventional therapy in acute heart failure patients.

DETAILED DESCRIPTION:
Study overview:

The purpose of this study is to evaluate whether ultrasound-guided decongestive therapy, guided by a focused thoracic ultrasound protocol combining echocardiography and lung ultrasound, could result in better decongestion and post-discharge prognosis without lengthening hospitalizations in hospitalized Acute Heart Failure patients.

Primary objectives:

To test whether ultrasound-guided therapy could result in reduced 6-month post-discharge mortality rates or re-hospitalization rates

Secondary objectives:

To test whether ultrassound-guided therapy could result in greater decongestion as defined by various congestion parameters, i.e. ultrasound-derived cardiac filling pressures on echocardiography, pulmonary congestion on lung ultrasound, reduction in natriuretic peptides and symptoms, fluid loss etc, and if this can be done without an increase in adverse events or and increase in length of hospitalizations.

Study Design and population:

ECHO-AHF is a non-blinded, randomized trial which will be conducted in 3-5 centers across Europe. Patients entering the ED between 8 am and 5 pm, monday to friady, and who fulfill study criteria will be enrolled and randomized in a 1:1-fashion

Inclusion criteria will consist of: Age 18 years or older and dyspnea at rest or orthophnea, BNP >400ng/l or a BNP >100ng/l AND signs of elevated LVEDP on echocardiography and multiple bilateral B-lines on LUS,. Dyspnea on excertion will not be sufficient for enrolment.

Exclusion criteria will consist of: Pulmonary fibrosis, Mental confusion, Chronic dialysis, Pregnancy/breastfeeding, Prisoners, Patient under involuntary treatment, Decision on study participation not made within 6 hours after receiving information regarding the study.

Estimated population size based on power calculation will be approximately 120 patients in total.

Investigational therapy in the treatment group:

Patients randomized to the treatment arm will receive ultrasound-guided therapy based on a focused ultrasound exam done on a daily basis except for saturdays and sundays, and their treatment will be intensified according to a pre-specified, guideline-based treatment protocol, if the daily ultrasound protocol finds them congestive. Patients in the control arm will receive guideline-based conventional decongestive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Multiple bilateral B-lines as a sign of interstitial syndrome on lung ultrasound
* Elevated natriuretic peptide level
* Signs of elevated LVEDP on echocardiography
* Dyspnea at rest or ortophnea

Exclusion Criteria:

* eGFR <25ml/min/1.73m2 or on dialysis
* Altered mental orientation
* Intubated
* Mitral stenosis or previous mitral valve procedure
* Chronic pulmonary parenchymal disease Pregnancy/breastfeeding
* Prisoners
* Patient under involuntary treatment
* Decision on study participation not made within 6 hours after receiving information regarding the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with re-hospitalization or death | 6-months, also 3-months will be analyzed
  post-discharge combined endpoint of re-hospitalization for acute heart failure or death due to any cause
Number of patients with re-hospitalization | 6-months, also 3-months will be analyzed
  Post-discharge re-hospitalization due to acute heart failure

SECONDARY OUTCOMES:
Number of patients with decongestion | during hospitalization
  Decongestion as measured by multiple congestion parameters, i.e. reduction in cardiac filling pressures and pulmonary congestion on ultrasound, fluid/weight loss, reduction in natriuretic peptides, symptom improvement, length of hospitalization, adverse events

IPD SHARING:
Plan to Share IPD: No